CLINICAL TRIAL: NCT04575870
Title: Return of Aspiration-Free Swallow After Laryngotracheal Anesthesia (LTA)
Brief Title: Return of Aspiration-Free Swallow After Laryngotracheal Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Blake Simpson, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005704
Record Dates: First submitted 2020-08-07; First posted 2020-10-05 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Swallowing, Air
MeSH Terms: conditions — Aerophagy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment Group 1: 90 min waiting period: Participants undergo their planned tracheobronchoscopy + 90 minute waiting period prior to modified functional endoscopic swallowing exam
  Interventions: Other: waiting period
- Treatment Group 2: 66 min waiting period: Participants undergo their planned tracheobronchoscopy + 66 minute waiting period prior to modified functional endoscopic swallowing exam
  Interventions: Other: waiting period
- Treatment Group 3: 46 min waiting period: Participants undergo their planned tracheobronchoscopy + 46 minute waiting period prior to modified functional endoscopic swallowing exam
  Interventions: Other: waiting period

INTERVENTIONS:
Other: waiting period — amount of time between clinical procedure and modified functional endoscopic exam of swallowing

SUMMARY:
Patients undergo laryngotracheal anesthesia (LTA) for a variety of in-office laryngology procedures. Prior to resolution of laryngeal sensory anesthesia, oral intake may predispose patients to aspiration. The purpose of this study is to objectively characterize a time period for return of aspiration-free swallow after LTA.

DETAILED DESCRIPTION:
Swallowing is a complex process involving coordination of multiple muscle groups. Sensation in the throat is very important for swallowing safely. Laryngotracheal anesthetic (LTA, or topical application of lidocaine anesthetic to larynx and trachea) is needed for a variety of in-office laryngology procedures, including examination of the air passage, or tracheobronchoscopy. This causes a temporary decrease in sensation that can affect swallow function and result in aspiration (passage of swallowed material into lungs instead of into esophagus and stomach). It is not known how long this effect lasts. It would be helpful to know this for counseling patients on when they can resume swallowing after a procedure. In general, most patients are advised to avoid eating/drinking for 90 minutes after their procedure to allow for sensation to return. To date, there has been no study characterizing the time required for return of aspiration-free swallow after LTA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability of patients to speak and understand English
* Ability for patients to consent for themselves
* Undergoing tracheobronchoscopy procedure for the treatment of airway stenosis
* Eating Assessment Tool (EAT-10) score ≤ 3

Exclusion Criteria:

* Age less than 18 years
* Patients unable or unwilling to provide informed consent
* Women who are pregnant
* History of abnormal swallowing evaluation, either videofluroscopic study of swallow or functional endoscopic evaluation of swallowing (FEES)
* History of medical condition affecting swallowing, such as

  * Neurodegenerative disorders: stroke, traumatic brain injury, dementia, motor neuron disease, myasthenia gravis, cerebral palsy, Gullain-Barre syndrome, poliomyelitis, myopathy, Parksonism, Huntingon's disease, progressive supranuclear palsy, Wilson's disease, vocal fold paralysis
  * Connective tissue disorders: polymyositis, dermatomyositis, progressive systemic sclerosis, Sjogren's disease, scleroderma
  * History of gastroesophageal tumor
  * History of gastroesophageal surgery
  * History of recent open central neck surgery (i.e., thyroidectomy, anterior cervical discectomy or fusion)
  * History of head and neck cancer
  * History of head and neck radiation therapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment for airway stenosis who present to the University of Alabama at Birmingham Voice Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Modified functional endoscopic exam of swallowing (FEES) | Up to 90 minutes
  A modified functional endoscopic exam of swallowing (FEES) is an examination where a small amount of water will be ingested. Each subject will perform about three water swallows. Water will be dyed with green food coloring to facilitate visualization, as is standard with the FEES procedure. If the water passes normally to the esophagus, this will be considered a pass; if the water is aspirated, this will be considered a fail.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Simpson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No